CLINICAL TRIAL: NCT01772550
Title: A Randomized Controlled Study to Determine Whether Smaller Gauge Fenestrated Catheters Are as Effective as Larger Gauge Non-fenestrated Catheters for Use in IV Contrast Enhanced CT Scans
Brief Title: Study of Effectiveness of Smaller Gauge Fenestrated Catheters for Use in IV Contrast Enhanced CT Scans
Acronym: ARCTR05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INF-11-ARCTR05
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Contrast Enhanced Computed Tomography
Keywords: CECT, catheter, contrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 Gauge BD Nexiva Diffusics (Experimental): During their routinely scheduled contrast-enhanced computed tomography procedure, subjects in this arm will receive IV contrast media injected via the fenestrated 20GA BD Nexiva Diffusics single port IV catheter (20GA x 1.00 inch).
  Interventions: Device: 20GA BD Nexiva Diffusics
- 18 Gauge Conventional Catheter (Active Comparator): During their routinely scheduled contrast-enhanced computed tomography procedure, subjects in this arm will receive IV contrast media injected via the non-fenestrated 18GA Conventional Catheter (18 GA x 1.25 inch Smiths Medical Jelco® IV Catheter).
  Interventions: Device: 18GA Conventional Catheter
- BD Nexiva Diffusics - Nonrandomized (Experimental): Subjects whose veins were not suitable for an 18 GA IV Catheter were assigned to this non-randomized arm. During their routinely scheduled CECT procedure, subjects receive IV contrast medium injected via the fenestrated 20GA BD Nexiva Diffusics single port IV catheter (20GA x 1.00 inch)
  Interventions: Device: 20GA BD Nexiva Diffusics

INTERVENTIONS:
Device: 20GA BD Nexiva Diffusics — The Inserter will have a single attempt on each arm (antecubital area) in which to insert the study catheter. If the catheter is not successfully inserted on the first attempt, the Inserter may make a second attempt in the contralateral arm.
  If the Inserter is unsuccessful in the second attempt, the subject is to be discontinued from the Study, and additional (non-Study) insertion attempts may be made according to facility policies.
  Other Names: 20G x 1 inch BD Nexiva™ Diffusics™ IV catheter (#383592)
  Arms: 20 Gauge BD Nexiva Diffusics; BD Nexiva Diffusics - Nonrandomized
Device: 18GA Conventional Catheter — The Inserter will have a single attempt on each arm (antecubital area) in which to insert the study catheter. If the catheter is not successfully inserted on the first attempt, the Inserter may make a second attempt in the contralateral arm.
  If after the first attempt, there is no vein in the contralateral arm that can accommodate an 18 gauge catheter, the subject is to be discontinued from the Study, and additional (non-Study) insertion attempts may be made according to facility policies.
  Other Names: 18G x 1.25 inch Smiths Medical Jelco® IV Catheter (cat#4055)
  Arms: 18 Gauge Conventional Catheter

SUMMARY:
The purpose of this study is to compare multidetector computed tomography (CT) image quality following peripheral venous high pressure injection of iodinated intravenous contrast media between a 20 gauge (GA) fenestrated, intravenous catheter (BD Nexiva™ Diffusics™) and an 18 GA non-fenestrated, intravenous catheter.

In the contrast enhanced CT procedure (CECT), a machine (power injector) is used to rapidly deliver contrast agent to an individual's circulatory system. The contrast allows for greater differentiation of tissues in images of the area of interest, affording a better opportunity to visually assess the area and hence make a more accurate diagnosis.

CECT often requires a high rate of contrast flow (≥ 5 mL/sec) through the IV catheter to provide sufficient contrast for an acceptable image. Typically an 18 GA IV catheter is required to achieve these high flow rates; however, often the patient does not have a vein that will accommodate this large size catheter. The BD Nexiva™ Diffusics™ IV catheter is designed to deliver a higher flow rate than a conventional catheter of the same gauge by incorporating fenestrations (small openings) near the tip of the catheter that allow fluid to exit the catheter in addition to that which normally exits through the main opening at the tip of the catheter.

DETAILED DESCRIPTION:
This is a prospective study performed in adult human subjects who have been referred for a CECT. The study will occur during a single visit. Once consented and enrolled, subjects whose antecubital veins can accommodate an 18 GA IV catheter (as assessed by the Inserter or designee of the PI), will be randomized to receive either a conventional 18 GA IV catheter (reference, control) or a 20 GA BD Nexiva™ Diffusics™ IV catheter (test). Subjects whose veins are not considered suitable for an 18 GA IV catheter will be placed in a non-randomized cohort for placement of a 20 GA BD Nexiva™ Diffusics™ IV catheter. Subjects will receive one (1) catheter for the study.

The primary objective of this study is to compare multidetector computed tomography (CT) image quality following peripheral venous high pressure injection of iodinated intravenous contrast media between a 20 GA fenestrated, intravenous catheter (BD Nexiva™ Diffusics™) and an 18 GA non-fenestrated, intravenous catheter. The 20 GA BD Nexiva™ Diffusics™ IV catheter will be considered non-inferior to conventional 18 GA IV catheters if the 95% upper bound for the difference in percentage of images of acceptable quality between the images acquired using the 18 GA IV catheters and the 20 GA BD Nexiva™ Diffusics™ IV catheters is less than 15%.

Study catheters will be inserted by appropriately licensed healthcare professionals (Inserters). Prior to enrollment, potential Inserters will be trained and qualified by the Sponsor on proper use of the BD Nexiva™ Diffusics™ IV catheter in both an artificial hand model and then in human patients. Inserters will then be expected to use the test product for a period of two (2) weeks, in order to gain familiarity with the product. Because BD Nexiva™ Diffusics™ IV catheters are not currently used in the Johns Hopkins Outpatient Center, the Sponsor will provide BD Nexiva™ Diffusics™ IV catheters for use during this training and familiarization period.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old at the time of enrollment,
* Must meet the investigational site's standard criteria for multi-detector Computed Tomography (CT),
* Per institutional protocol, the ordered scan must require a flow rate of 5.0-7.0 mL/sec (inclusive) for Visipaque 320 or 5.0-7.5 mL/sec (inclusive) for Omnipaque350 warmed to 35°C,
* The planned catheter insertion site must be located in the antecubital area,
* Must require any of the following multi-detector CT procedures: CT angiogram,CT pancreas,CT liver, CT kidney, Cardiac CT,
* Must be willing and able to provide informed consent,
* Must be able to read, write, and follow instructions in English,
* Must be able to accommodate a 20 G x 1.00 inch IV catheter,

Exclusion Criteria:

* Preexisting IV catheter or contrast-compatible port in place suitable for power injection with the intent to be used for contrast enhanced CT,
* Subjects who have reported an adverse reaction that precludes use of iodine-based contrast media,
* Subjects who have had a prior extravasation event involving solutions considered irritants or vesicants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Fishman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from those referred to the Johns Hopkins Outpatient Center for contrast enhanced computed tomography, or CECT. Subjects were recruited in January and February of 2013.
  The Overall Study table summarizes the number of subjects that Started and Completed in each Reporting Group, including the type of CECT procedure.
Pre-assignment Details: Subjects whose veins were determined to be unable to accommodate an 18 GA IV catheter, but that could accommodate a 20 GA IV catheter, were not randomized but were assigned to receive the 20 GA BD Nexiva™ Diffusics™ IV catheter (non-randomized cohort).
Groups:
- 20 GA BD Nexiva Diffusics - Randomized: During their routinely scheduled CECT procedure, subjects receive IV contrast medium injected via the 20 GA fenestrated BD Nexiva Diffusics single port IV catheter
- 18 GA Conventional Catheter - Randomized: During their routinely scheduled CECT procedure, subjects receive IV contrast medium injected via the non-fenestrated 18GA x 1.25 inch Smiths Medical Jelco IV catheter
- 20 GA BD Nexiva Diffusics - Nonrandomized: Subjects whose veins are not suitable for an 18GA IV catheter will be assigned to this non-randomized arm. During their routinely scheduled CECT procedure, subjects receive IV contrast medium injected via the 20GA fenestrated BD Nexiva Diffusics single port IV catheter
Period: Overall Study
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Started | 102 | 103 | 33
CT Pancreas | 40 | 36 | 8
CT Angiogram | 24 | 25 | 4
CT Liver | 18 | 14 | 8
CT Kidney | 12 | 19 | 6
CT Cardiac | 7 | 7 | 1
Completed | 101 | 102 | 27
Not Completed | 1 | 1 | 6
Not completed — Unable to insert IV in antecubital vein | 1 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized | Total
Number analyzed (Participants) | 102 | 103 | 33 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.9) | 60.0 (13.6) | 58.8 (12.3) | 60.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 37 | 20 | 102
  Male | 57 | 66 | 13 | 136

OUTCOME MEASURES:

1. Primary Outcome: Acceptable Image Quality
Description: Study images were assessed by a US board-certified radiologist to determine whether the image is of acceptable quality. The radiologist was not informed of the study device used for the injection that produced the image under evaluation. Subjective image quality assessment for acceptability was determined by:
  * The report of the reading radiologist in the section of the report where the radiologist indicates if the image is acceptable or not. The absence of a comment in this section will be interpreted as acceptable, and,
  * the assessment of an independent single second reader (such as the subinvestigator or research radiologist) blinded to the reading radiologist's report and the infusion catheter type.
  In the case of a non-concurrence, the Principal Investigator assessed the image and his or her assessment had final authority.
Time Frame: at the time of image assessment
Population: One subject randomized to the 18 GA conventional catheter was excluded from the per-protocol analysis. Due to catheter placement, the required minimum flow rate of 5 mL/sec could not be achieved; contrast was administered at 4.5 mL/sec.
Measure: Number; unit: percentage of participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 27
percentage of participants | 100 | 100 | 100
Statistical Analysis 1: Comparison: 20 GA BD Nexiva Diffusics - Randomized vs 18 GA Conventional Catheter - Randomized; Only the percent of acceptable image quality from the randomized test and reference catheter groups were considered for this statistical analysis. If C is the percentage of acceptable quality images with the control catheter, and D is the percentage of images of acceptable quality with the evaluation catheter, and the non-inferiority criteria is 15%, the hypotheses to be tested are as follows: H0: C - D > or = 15%; H1: C - D < 15%; Test type: Non-Inferiority or Equivalence — A 95% upper confidence bound for the observed difference in percentages of images with acceptable quality between the control catheter and evaluation catheter was calculated using the Score method. The 20 G BD Nexiva™ Diffusics™ can be considered non-inferior for acceptable image quality if this 95% upper confidence bound is smaller than 15% (i.e. C - D < 15% with 95% confidence). The non-inferiority margin was 15%; Risk Difference (RD) = 0, 95% CI 1-sided [upper limit 2.6] — The difference in percent of acceptable image quality is used as an estimate. The Score method was used to estimate the upper 95% confidence limit

2. Secondary Outcome: Abdomen CT - Average Hounsfield Units as a Measure of Aortic Contrast Delivery and Enhancement in Randomized Subjects
Description: Objective image quality assessment was performed by a board-certified Research Radiologist, by measuring the post-contrast aortic attenuation in Hounsfield Units (HU) at either the aortic arch if chest is imaged or the diaphragmatic crus and above the aortic bifurcation or on the most inferior image on the arterial phase. Hounsfield units within the proximal and distal aorta were recorded for each subject image reviewed. The average number of HU for each group in the Study are reported descriptively; formal acceptance criteria for this objective are not specified.
Time Frame: at the time of image assessment
Population: 126 subjects had HU measurements available from abdominal CT imaging.
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized
Number analyzed (Participants) | 63 | 63
Hounsfield Units | 400.9 (69.8) | 402.5 (91.5)

3. Secondary Outcome: Chest CT - Average Hounsfield Units as a Measure of Aortic Contrast Delivery and Enhancement in Subjects Whose Veins Could Accommodate an 18 GA IV Catheter (Randomized Subjects)
Description: as for outcome 2
Time Frame: at the time of image assessment
Population: 20 subjects had HU measurements available from thoracic CT imaging.
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized
Number analyzed (Participants) | 10 | 10
Hounsfield Units | 428.9 (76.9) | 402.2 (87.2)

4. Secondary Outcome: Complete Chest and Abdomen CT - Average Hounsfield Units as a Measure of Aortic Contrast Delivery and Enhancement in Subjects Whose Veins Could Accommodate an 18 GA IV Catheter (Randomized Subjects)
Description: as for outcome 2
Time Frame: at the time of image assessment
Population: 54 subjects had HU measurements available from complete chest and abdomen CT imaging.
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized
Number analyzed (Participants) | 27 | 27
Hounsfield Units | 373.2 (68.9) | 387.7 (71.7)

5. Secondary Outcome: Maximum Flow Rate
Description: Maximum flow rate guidelines provided in the BD Nexiva Diffusics Instructions for Use were to be followed. The maximum flow rate (milliliters per second, or mL/sec) utilized was recorded by the Radiology Technician immediately following the power injection of iodinated intravenous contrast media. Results are descriptively summarized; no formal acceptance criteria were specified by the protocol.
Time Frame: immediately after power injection
Population: One subject randomized to the 18 GA conventional IV was excluded from the analysis as the required minimum flow rate could not be achieved due to IV placement. Non-randomized flow rate analysis only includes subjects who completed successful contrast delivery; one subject with extravasation upon delivery was discontinued and is not included.
Measure: Mean (Standard Deviation); unit: mL/second
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 27
mL/second | 5.58 (0.49) | 5.74 (0.66) | 5.46 (0.44)

6. Secondary Outcome: Catheter Insertion Success
Description: Insertion is successful when the catheter can be flushed or infused to demonstrate patency, and there is no inadvertent administration of a solution or medication into the tissue surrounding the IV catheter.
  The number of participants with successfully inserted catheters after the first or second insertion attempt is reported. The clinician inserting the IV catheter made a clinical judgement as to whether the catheter was successfully placed; the protocol did not define more specific criteria. Catheter insertion success rates were determined from each IV insertion attempted in the Study.
Time Frame: immediately after catheter insertion
Population: All subjects for whom an insertion was attempted are included in the analysis for insertion success. This includes some subjects that did not go on to complete the study.
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 102 | 103 | 33
participants
  Success with first insertion attempt | 96 | 100 | 20
  Success with second attempt | 5 | 2 | 8
  Unsuccessful after second attempt | 1 | 1 | 5

7. Secondary Outcome: Extravasation of Contrast Media
Description: The number of subjects who experienced injections with extravasation of contrast media is reported.
Time Frame: upon contrast injection
Population: One subject randomized to the 18 GA IV was excluded from the per-protocol analysis as minimum flow rate could not be achieved. Non-randomized group analysis includes 1 subject with media extravasation with first study IV (adverse event). Subject was discontinued and not included in primary outcomes analysis.
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 28
participants | 0 | 0 | 1

8. Secondary Outcome: Automatic Injection Shutoff
Description: The number of subjects who experienced injections with automatic injection shutoff is reported. Immediately after the power injection, the injection technician recorded whether or not an automatic injection shutoff occurred.
Time Frame: immediately after contrast injection
Population: One subject randomized to the 18 GA conventional IV was excluded from the analysis as the required minimum flow rate could not be achieved due to IV placement. Non-randomized group analysis includes 1 subject with media extravasation with first study IV (adverse event). Subject was discontinued and not included in primary outcomes analysis.
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 28
participants | 0 | 0 | 0

9. Secondary Outcome: High Pressure Alarm
Description: The number of subjects who experienced injections with activation of the high pressure alarm is reported. Immediately following the power injection, the clinician performing the power injection recorded whether or not the high pressure alarm sounded.
Time Frame: immediately after contrast injection
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 28
participants | 0 | 1 | 1

10. Secondary Outcome: Catheter Dislodgement
Description: The number of subjects who experienced partial or complete dislodgement of the catheter from the subject prior to power injection procedure completion is reported. The information about the IV catheter was collected by a clinically qualified study staff member (e.g., the Principal or sub-Investigator, or Study Coordinator) after the power injection.
Time Frame: Immediately following power injection
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 28
participants | 0 | 0 | 0

11. Secondary Outcome: Catheter Transfixation
Description: The number of subjects who experienced catheter transfixation (the IV penetrating the opposite wall of the vein) is reported. This information was collected by a clinically qualified study staff member (e.g., the Principal or sub-Investigator, or Study Coordinator) after the power injection.
Time Frame: immediately after power injection
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 28
participants | 0 | 0 | 0

12. Secondary Outcome: Catheter Integrity Failure
Description: Catheter integrity failure generally refers to any portion of the device breaking or malfunctioning so that its proper function is no longer assured. In this study, the most relevant catheter integrity failures to be assessed were fluid leakage, tubing rupture, or tubing separation from the hub.
  The number of subjects who experienced injections with a catheter integrity failure during injection is reported. The information about the IV catheter was collected by a clinically qualified study staff member (e.g., the Principal or sub-Investigator, or Study Coordinator) after the power injection.
Time Frame: immediately after power injection
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Number analyzed (Participants) | 101 | 101 | 28
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 20 GA BD Nexiva Diffusics - Randomized | 18 GA Conventional Catheter - Randomized | 20 GA BD Nexiva Diffusics - Nonrandomized
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/103 | 0/33
Other Adverse Events (participants affected / at risk) | 0/102 | 0/103 | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 GA BD Nexiva Diffusics - Randomized (N=102) | 18 GA Conventional Catheter - Randomized (N=103) | 20 GA BD Nexiva Diffusics - Nonrandomized (N=33)
Extravasation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less